CLINICAL TRIAL: NCT02293148
Title: A Two-part Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a High, Single Oral Dose of GSK1278863 (Part A), and a Randomized, Single-blind, Placebo- and Positive-controlled, Four-way Crossover Study to Assess the Effect of Single, Oral Dose of GSK1278863 on Cardiac Repolarization (Part B) in Healthy Volunteers
Brief Title: Single Dose, Pharmacokinetic, Safety, Tolerability and QTc Study of GSK1278863 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113635
Record Dates: First submitted 2014-11-03; First posted 2014-11-18 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Anaemia
Keywords: Prolyl hydroxylase inhibitor; GSK1278863; Anemia; QTc; erythropoiesis stimulating agent
MeSH Terms: conditions — Anemia | interventions — GSK1278863; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1278863 (Part A) (Experimental): All subjects will receive a single, oral 500 mg dose of GSK1278863 on Day 1 administered as 5 x 100 mg tablets of GSK1278863. Additional doses/cohorts may be added depending upon the emerging safety, tolerability, pharmacokinetic and/or pharmacodynamics findings at the 500 mg dose level in Part A
  Interventions: Drug: GSK1278863 500 mg
- GSK1278863 (75 mg/500 mg)/Moxifloxacin 400 mg/Placebo (Part B) (Experimental): Subjects will be assigned to one of four treatment sequences (A-1 x Moxifloxacin placebo tablet, 3 x 25 mg tablets of GSK1278863, 2 x GSK1278863 matched placebo; B-1 x Moxifloxacin placebo tablet, 5 x 100 mg tablets of GSK1278863; C-1 x Moxifloxacin placebo tablet, 5 x GSK1278863 matched placebo tablets; D-1 x 400 mg Moxifloxacin tablet, 5 x GSK1278863 matched placebo tablets) (ABDC, BCAD, CDBA, DACB) in accordance with the randomization schedule
  Interventions: Drug: GSK1278863 75 mg; Drug: GSK1278863 500 mg; Drug: Moxifloxacin 400 mg; Drug: Placebo matching GSK1278863; Drug: Placebo matching Moxifloxacin

INTERVENTIONS:
Drug: GSK1278863 75 mg — A round, biconvex, white film coated tablet available in two doses (25 and 100 mg)
  Arms: GSK1278863 (75 mg/500 mg)/Moxifloxacin 400 mg/Placebo (Part B)
Drug: GSK1278863 500 mg — A round, biconvex, white film coated tablet available in two doses (25 and 100 mg)
Drug: Moxifloxacin 400 mg — Oblong, dull red, film-coated, convex tablets with M400 on one side
  Arms: GSK1278863 (75 mg/500 mg)/Moxifloxacin 400 mg/Placebo (Part B)
Drug: Placebo matching GSK1278863 — A round, biconvex, white film coated tablet as matching placebo for GSK1278863
  Arms: GSK1278863 (75 mg/500 mg)/Moxifloxacin 400 mg/Placebo (Part B)
Drug: Placebo matching Moxifloxacin — Capsule shaped white film coated tablet as matching placebo for Moxifloxacin
  Arms: GSK1278863 (75 mg/500 mg)/Moxifloxacin 400 mg/Placebo (Part B)

SUMMARY:
This study is being performed to comply with regulatory requirements that all new non-antiarrhythmic drugs must be assessed for potential effects on cardiac repolarization through electrocardiographic evaluation in a 'Thorough QT/ Corrected QT interval (TQT)' study. This will be a two part study, Part A will be an open-label, single oral dose study design in order to evaluate the pharmacokinetics, safety and tolerability of a 500 milligram (mg) dose of GSK1278863 and Part B will be a single-blind, randomized, placebo-controlled, single, oral dose, four-way crossover study design. Parts A and B will be conducted in healthy adult subjects with 12-lead electrocardiograms (ECGs), clinical laboratory safety tests, vital sign measurements, physical examinations, adverse event reports, and pharmacokinetic samples collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are between 18 and 45 years and of age, inclusive at the time of signing the informed consent form
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring obtained at the Screening visit.

The determination of clinical significance will be made by the Investigator and the GlaxoSmithKline (GSK) Medical Monitor and will require that the finding is unlikely to introduce additional risk factors or interfere with the study procedures, or the integrity of the study

* Hemoglobin values at screening greater than the lower limit of the laboratory reference range and less than or equal to 16.0 gram (g)/decilitre (dL) for males and less than or equal to 14.0 g/dL for females
* No significant abnormality on 12-lead ECG at screening, including the following specific requirements:

Ventricular rate >= 40 beats per minute; PR interval <= 210milliseconds (msec); Q waves < 30msec (up to 50msec permitted in lead III only); QRS interval to be >= 60msec and < 120msec; The waveforms must enable the QT interval to be clearly defined; QTcF interval must be < 450msec.

* Body weight >= 50 kilograms (kg) and body mass index (BMI) within the range 19-29.9 kg/meter square (m^2) (inclusive).
* Female and Male:

Female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

* Non-reproductive potential defined as:
* Pre-menopausal females with one of the following:
* Documented tubal ligation
* Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion
* Hysterectomy
* Documented Bilateral Oophorectomy
* Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases, a blood sample with simultaneous follicle stimulating hormone (FSH) 23.0-116.3 International Units (IU)/Litre (L) and estradiol <=10 picograms (pg)/millilitre (mL) (or<=37 Picomoles (pmol)/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment
* Reproductive potential and agrees to follow the contraception requirement for female subjects from 30 days prior to the first dose of study treatment and until at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer after the last dose of study treatment and completion of the follow-up visit
* Capable of giving signed informed consent and includes compliance with the requirements and restrictions listed in the consent form and in this protocol

Exclusion Criteria:

* Hypertensive (diastolic BP >90 millimetres of mercury [mmHg] or systolic BP >140 mmHg) at screening
* A supine mean heart rate outside the range 50-100 beats per minute (bpm) at screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin >1.5x Upper Limit of Normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* History or presence of any medically significant disease, or any disorder that would introduce additional risk or interfere with the study procedures or outcome. In particular, a family history of QT prolongation, of early or sudden cardiac death or of early cardiovascular disease

NOTES:

* The QTc is the QTcF interval
* The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial
* Serum calcium, magnesium or potassium levels outside the normal reference range
* History of deep vein thrombosis, stroke, transient ischemic attack, pulmonary embolism or other thrombosis related condition within the last five years
* History of myocardial infarction or acute coronary syndrome
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, and/or hepatic function that could interfere with the absorption, metabolism, and/or excretion of GSK1278863. Examples of conditions that could interfere with normal gastrointestinal anatomy or motility include gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, or celiac sprue
* Evidence of active peptic, duodenal or esophageal ulcer disease at Screening OR history of clinically significant gastrointestinal bleeding
* Subjects with chronic inflammatory joint disease (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis)
* Subjects with a history of pulmonary artery hypertension
* Subjects with heart failure, as defined by the New York Heart Association (NYHA) functional classification system, including known right heart failure
* Subjects with a history of malignancy within the prior five years, who are receiving treatment for cancer, or who have a strong family history of cancer (e.g., familial cancer disorders); with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated prior to screening through Day -1 (Randomization)
* History of proliferative vascular eye disease (e.g., choroidal or retinal disease, such as neovascular age-related macular degeneration, proliferative diabetic retinopathy or macular edema)
* Subjects must abstain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements) except occasional usage of acetaminophen, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment until completion of the follow-up visit, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study medications)
* History of regular alcohol consumption within 6 months of the study defined as:

An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits

* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products prior to screening
* History of regular use within 6 months of the study of tobacco- or nicotine-containing products
* History of drug abuse or dependence within 6 months of the study
* History of sensitivity to GSK1278863, or its components thereof, a history of sensitivity to quinolone antibiotics or components thereof, or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation
* Consumption of red wine, grapefruit (juice), blood orange (juice), star fruit, onions, kale, broccoli, green beans, or apples from 7 days prior to the first dose of study treatment until the Follow-up visit, unless in the opinion of the Investigator and GSK Medical Monitor this will not interfere with the study procedures and compromise subject safety
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency)
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines
* A positive test for Human Immunodeficiency Virus antibody
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the study treatment (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unwillingness or inability to follow the procedures outlined in the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2015-03-10 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters for GSK1278863 and its metabolites for Part A | Pre Dose, 0.25hour (h), 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 18h, and 24h post dose in each treatment period
  Plasma concentrations of GSK1278863 and its metabolites (GSK2391220 [M2], GSK2506104 [M3], GSK2487818 [M4], GSK2506102 [M5], GSK2531398 [M6], and GSK2531401 [M13]) and derived pharmacokinetic parameters including maximum observed concentration (Cmax), Time of occurrence of Cmax (tmax), Area under the concentration-time curve (AUC)
Change from baseline in QT duration corrected for heart rate by Fridericia's formula (QTcF) interval for Part B | At each treatment period (there are 4 periods) up to 24 hours
  Change from baseline in QTcF interval at each time-point (average of at least three 12-lead Holter ECG replicates per time-point (Pre-dose, Day 1 [0.25h, 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 18h] and 24h) for 75 and 500 mg dose of GSK1278863 as compared with time-matched placebo
Assessment of 12-lead ECG for Part A | Up to Week 3
  12-lead ECGs will be obtained at each time-point
Assessment of Vital Signs for Part A | Up to Week 3
  Vital Signs includes. temperature, systolic and diastolic blood pressure (BP) and pulse
Number of participants with Adverse Events (AE) for Part A | Up to Week 3
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Assessment of Clinical Laboratory Tests for Part A | Up to Week 3
  Clinical Laboratory Tests includes Hematology, Clinical Chemistry and Urinalysis

SECONDARY OUTCOMES:
Change from baseline in QT duration corrected for heart rate by Bazett's formula (QTcB), heart rate (HR), PR, QRS, and QT interval corrected for heart rate (QTci/QTciL interval) for GSK1278863 for Part B | Up to Week 9
  Change from baseline in QTcB, HR, PR, QRS and QTci/QTciL interval at each time-point (average of at least 3 12-lead Holter ECG replicates per time-point) for 75 mg and 500 mg dose of GSK1278863 as compared with time-matched placebo
Change from baseline in QTcB, HR, PR, QRS, and QTci/QTciL interval for moxifloxacin for Part B | Up to Week 9
  Change from baseline in QTcF, QTcB, and QTci/QTciL interval at each time-point (average of at least 3 12-lead Holter ECG replicates per time-point) for 400 mg dose of moxifloxacin as compared with time-matched placebo
Composite of PK parameters for GSK1278863, its metabolites and moxifloxacin for Part B | Pre-dose, 0.25h, 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 18h, and 24h in each treatment period of part B
  Plasma concentrations of GSK1278863, and its metabolites GSK2391220 (M2), GSK2506104 (M3), GSK2487818 (M4), GSK2506102 (M5), GSK2531398 (M6), and GSK2531401 (M13), moxifloxacin, and derived pharmacokinetic parameters including Cmax, tmax, AUC
Maximal change from baseline in ECG parameters for Part B | Up to Week 9
  Maximal change from baseline in ECG parameters for QTcF and QTcB
Change from baseline for other ECG parameters for Part B | Up to Week 9
  Change from baseline at each time-point for other cardiac electrophysiological parameters: QT, QRS, RR, PR and ventricular rate
Change in QTc Cmax for Part B | Up to Week 9
  Evaluate the slope of the relationship and the predicted median (90% confidence interval [CI]) value of change in QTc Cmax following therapeutic doses
Assessment of Vital Signs for Part B | Up to Week 9
  Vital Signs includes. temperature, systolic and diastolic blood pressure and pulse
Number of participants with Adverse Events in Part B | Up to Week 9
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Assessment of Clinical Laboratory Tests for Part B | Up to Week 9
  Clinical Laboratory Tests includes Hematology, Clinical Chemistry and Urinalysis
ECG assessment as a safety measure in Part B | Up to Week 9
  Triplicate 12-lead ECGs will be obtained at each time-point (Day -1, Pre-dose, Day 1 [0.25h, 0.5h, 1h, 2h, 3h, 4h, 5h, 6h, 8h, 12h, 18h], Day 2 [24h])during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: Results for study 113635 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113635?search=study&study_ids=113635#rs